CLINICAL TRIAL: NCT05297786
Title: Prevention of Dialysis-Induced Hypotension by Inhibiting Plasma Kallikrein
Brief Title: Hemodialysis.-Induced Hypotension Therapy for End Stage Kidney Disease
Acronym: Hinder
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Jorge Gamboa, Research Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 210633
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Hemodialysis Complication; Hypotension of Hemodialysis
MeSH Terms: interventions — lanadelumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lanadelumab (Experimental): Subjects will receive lanadelumab (300 mg) subcutaneously at the beginning of the study and 14 days later
  Interventions: Drug: Lanadelumab Injection [Takhzyro]
- Placebo (Placebo Comparator): Subjects will receive placebo subcutaneously at the beginning of the study and 14 days later
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lanadelumab Injection [Takhzyro] — Lanadelumab 300 mg subcutaneous injection
  Arms: Lanadelumab
Drug: Placebo — Placebo injection
  Arms: Placebo

SUMMARY:
Bradykinin is a potent vasodilator that is formed by the activation of the kallikrein-kinin system. We and others have shown that bradykinin increased during hemodialysis; however, the role of bradykinin in dialysis-induced hypotension (DIH) has not been evaluated. Preliminary results from a pilot clinical trial showed that bradykinin B2 receptor blockade with icatibant prevents excessive blood pressure during hemodialysis. Thus, in this study, we will test the overarching hypothesis that blockade plasma kallikrein with lanadelumab would ameliorate the reduction of blood pressure during hemodialysis in patients who are prone to DIH. For this purpose, we will conduct a parallel arm, double-blind placebo-controlled trial, using lanadelumab to evaluate the occurrence of

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 to 85 years
* On thrice-weekly hemodialysis for at least six months
* Clinically stable, adequately dialyzed (single-pool Kt/V > 1.2), with polysulphone membrane for at least three consecutive months before the study
* Subjects with pre-dialytic systolic blood pressure between 110 and 170 mmHg.
* Subjects with a reduction of systolic blood pressure during hemodialysis equal to or greater than 30 mmHg, with associated symptoms such as nausea, vomiting, muscle cramps, dizziness, or anxiety.
* Hypotensive episodes should occur four times or more in four weeks (12 hemodialysis sessions).

Exclusion Criteria:

* Subjects with intradialytic hypotension that require the use of pharmacological intervention such as midodrine or vasopressin
* Subjects with pre-dialytic systolic blood pressure greater than 170 mmHg or diastolic blood pressure greater than 110 mmHg
* History of myocardial infarction or cerebrovascular event within 3 months
* History of serious hemorrhage (including cerebral hemorrhage) in the past 6 months
* Advanced liver disease
* Ejection fraction less than 30%
* Anticipated live donor kidney transplant
* A history of poor adherence to hemodialysis or medical regimen
* Severe anemia (hemoglobin less than 8 g/dl) requiring blood transfusions
* Use of immunosuppressive drugs within one month before study enrollment
* Active connective tissue disease
* History of acute infections disease within one month before study enrollment
* Inability to provide consent
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2026-01-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- Lanadelumab: Patients received 300 mg of lanadelumab subcutaneously on day 0 (the start of the study) and again on day 14
- Placebo: Patients received a placebo injection subcutaneously on day 0 (the start of the study) and again on day 14.
Period: Overall Study
Arm/Group | Lanadelumab | Placebo
Started | 14 | 14
Completed | 9 (Patients were enrolled, randomized, but do not received any study treatment) | 12 (Two patients received the first dose of study drug but not the second dose)
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Renal transplantation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lanadelumab | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (15.1) | 58.1 (13.9) | 59.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 10 | 21
  White | 3 | 3 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure During Hemodialysis
Description: Systolic blood pressure pre and post hemodialysis at baseline and at the end of the study
Time Frame: From the initiation of study until the end (week 6)
Population: Two patients in the placebo arm dropped after receiving the first dose of the study drug
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lanadelumab | Placebo
Number analyzed (Participants) | 9 | 14
mmHg
  Baseline-Pre hemodialysis | 155.9 (36.3) | 155.1 (28.8)
  Baseline-Post hemodialysis | 136.4 (26.8) | 126. (18.3)
  Six-weeks-Pre hemodialysis: number analyzed (Participants) | 9 | 12
  Six-weeks-Pre hemodialysis | 136.4 (18.5) | 141.5 (22.5)
  Six-weeks-Post hemodialysis: number analyzed (Participants) | 9 | 12
  Six-weeks-Post hemodialysis | 131.2 (15.8) | 119.0 (11.2)

2. Secondary Outcome: Hypotensive Episodes
Description: Number of hypotensive episodes during hemodialysis after the second week of treatment
Time Frame: From the second week of the study until the end (week 6)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Lanadelumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/9
Other Adverse Events (participants affected / at risk) | 4/14 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanadelumab (N=14) | Placebo (N=9)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) — Patient required hospitalization due to symptomatic bradicardia
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 2 (2) — Upper gastrointestinal bleeding
Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Rectal bleeding
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanadelumab (N=14) | Placebo (N=9)
Arterio-venous fistula occlusion (Vascular disorders) | 1 (1) | 0 (0)
Nausea or vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Headche (Nervous system disorders) | 2 (2) | 0 (0)
Menstrual cramps (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Swollen lips (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Dorsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT05297786/Prot_SAP_000.pdf